CLINICAL TRIAL: NCT03584672
Title: The Reliability, Validity, and Responsiveness of the Static Balance Test in Patients With Multiple Sclerosis.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fatih Söke, Research Assistant, Gazi University
Other Study IDs: 322
Record Dates: First submitted 2018-06-30; First posted 2018-07-12 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Static Balance Test; Balance; Reliability; Validity
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Multiple Sclerosis: Patients with Multiple Sclerosis (Expanded Disability Status Scale (EDSS) score < 7)
  Interventions: Other: Static Balance Test; Other: Berg Balance Scale; Other: Timed Up an Go Test; Other: Four Square Step Test; Other: Functional Reach Test; Other: One-leg Stance Test
- Healthy Controls: Healthy people
  Interventions: Other: Static Balance Test

INTERVENTIONS:
Other: Static Balance Test — Balance control is assessed by the Static Balance Test.
Other: Berg Balance Scale — Functional balance is assessed by the Berg Balance Scale.
  Groups: Patients with Multiple Sclerosis
Other: Timed Up an Go Test — Functional mobility is assessed by the Timed Up and Go test.
  Groups: Patients with Multiple Sclerosis
Other: Four Square Step Test — Dynamic balance is assessed by the Four Square Step Test.
  Groups: Patients with Multiple Sclerosis
Other: Functional Reach Test — Limits of stability is assessed by the Functional Reach Test.
  Groups: Patients with Multiple Sclerosis
Other: One-leg Stance Test — Postural steadiness is assessed by the One-leg Stance Test.
  Groups: Patients with Multiple Sclerosis

SUMMARY:
The aim of the study is to investigate reliability, validity, and responsiveness of the Static Balance Test in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
At baseline, the Static Balance Test, Berg Balance Scale, Timed Up and Go test, Functional Reach Test, Four Square Step Test, and One-legged Stance Test is applied to the Multiple Sclerosis group. The Static Balance Test is repeated after seven days from the first application in patients with Multiple Sclerosis. Healthy controls are going to perform only the Static Balance Test.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years,
* neurologist-diagnosed Multiple Sclerosis,
* Expanded Disability Status Scale (EDSS) score < 7,
* able to walk 10 m with or without aids,
* no MS exacerbation within the last 2 months,
* use of stable medication in the last 2 months,

Exclusion Criteria:

* other neurologic disorder,
* Pregnancy,
* orhopedic problems iaffecting gait and stance,
* visual, auditory, orientational problems that could affect study results,
* Cardiovascular, pulmonary, and humoral disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Sclerosis who apply to Gazi University, Department of Physiotherapy and Rehabilitation will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-08-05 (Estimated); Primary Completion 2018-08-20 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
Static Balance Test | 5 minutes
  The Static Balance Test is used to assess balance control. The Static Balance Test, consists of five posture-holding tasks (sitting, stride standing, close standing, one-foot standing on the unparalyzed leg, and one-foot standing on the paralyzed leg). Four grades, 1-4, are used to judge the ability of patients to hold these postures. The grade at which a subject is rated on a task is taken as the score for that task.
  Hence, the minimum Static Balance Test score is 5, and the maximum is 20. A higher score indicates better balance.

SECONDARY OUTCOMES:
Berg Balance Scale | 15 minutes
  Functional balance is assessed by using the Berg Balance Scale. During the test, participants are asked to perform 14 tasks frequently used in daily life activities. Each item is scored between 0 (unable to perform the task) and 4 (task is performed independently) according to the ability of the person while performing the task. The highest possible score is 56 points. A higher score indicates better balance.
Timed Up and Go Test | 1 minutes
  Functional mobility is assessed by using the timed up and go test. The timed up and go test measures the time that a patient needs to stand up from a chair, walk a 3-m distance, come back and sit back on the chair. A lower score indicates better functional mobility.
Four Square Step Test | 1 minutes
  The Four Square Step Test measures dynamic balance and clinically assesses the person's ability to step over objects forward, sideways, and backward. A square was formed by 4 canes resting flat on the floor. The participants were instructed to try and complete the sequence as fast as possible without touching the canes with both feet, making contact with the floor in each square. A lower score indicates better dynamic balance.
One-leg Stance Test | 5 minutes
  The clinical test of One-leg Stance Test assesses postural steadiness in a static position by a quantitative measurement i.e. the number of seconds a person can maintain the One-leg Stance Test position, thus implying that better postural steadiness would allow for longer standing on one leg.
Functional Reach Test | 30 seconds
  The Functional Reach Test assesses balance by measuring the limits while the patient reaches forwards as far as possible, having the arms in 90° flexion and without lifting the heels off the floor. A higher score indicates better limits of stability.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Söke, Principal Investigator — Gazi University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McConvey J, Bennett SE. Reliability of the Dynamic Gait Index in individuals with multiple sclerosis. Arch Phys Med Rehabil. 2005 Jan;86(1):130-3. doi: 10.1016/j.apmr.2003.11.033. PMID 15641003
- [Background] Gijbels D, Alders G, Van Hoof E, Charlier C, Roelants M, Broekmans T, Eijnde BO, Feys P. Predicting habitual walking performance in multiple sclerosis: relevance of capacity and self-report measures. Mult Scler. 2010 May;16(5):618-26. doi: 10.1177/1352458510361357. Epub 2010 Mar 5. PMID 20207785
- [Background] Matsuda PN, Shumway-Cook A, Bamer AM, Johnson SL, Amtmann D, Kraft GH. Falls in multiple sclerosis. PM R. 2011 Jul;3(7):624-32; quiz 632. doi: 10.1016/j.pmrj.2011.04.015. PMID 21777861
- [Background] Suzuki M, Fujisawa H, Machida Y, Minakata S. Relationship between the Berg Balance Scale and Static Balance Test in Hemiplegic Patients with Stroke. J Phys Ther Sci. 2013 Aug;25(8):1043-9. doi: 10.1589/jpts.25.1043. Epub 2013 Sep 20. PMID 24259912
- [Background] Cattaneo D, Regola A, Meotti M. Validity of six balance disorders scales in persons with multiple sclerosis. Disabil Rehabil. 2006 Jun 30;28(12):789-95. doi: 10.1080/09638280500404289. PMID 16754576